CLINICAL TRIAL: NCT07038330
Title: POSTOPERATIVE SUCROSOMIAL IRON IN HEART SURGERY: DOSE FINDING PROSPECTIVE STUDY (SideralDose)
Brief Title: DOSE FINDING PROSPECTIVE ANALYSIS AFTER HEART SURGERY for Sucrosomial Iron
Acronym: SideralDose
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cardiochirurgia E.H. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SideralDose
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Anemia
Keywords: Sucrosomial Iron; Oral Iron; Post Cardiac Surgery Rehabilitation
MeSH Terms: conditions — Anemia | interventions — sucrosomial iron

STUDY DESIGN:
Intervention Model Description: 1:1:1 randomization, one month administration,. two months follow up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 30mg (Experimental): 1 cp (30mg) per day of Sucrosomial Iron
  Interventions: Drug: Sucrosomial Iron
- 60mg (Experimental): 2 cp (60mg) per day of Sucrosomial Iron
  Interventions: Drug: Sucrosomial Iron
- 120mg (Experimental): 4 cp (120mg) per day of Sucrosomial Iron
  Interventions: Drug: Sucrosomial Iron

INTERVENTIONS:
Drug: Sucrosomial Iron — Sideral Forte, Italian market formulation of Sucrosomila Iron 30mg per cp

SUMMARY:
Randomization to different doses of Sucrosomial Iron for one moth after discharge to rehab after heart surgery to assess if more iron grants a faster recovery or not

DETAILED DESCRIPTION:
Evaluation of the efficacy of short-term sucrosomial iron treatment in patients undergoing cardiac surgery and subsequently transferred to rehabilitation, measured in terms of increase in hemoglobin values and restoration of martial blood parameters, administering doses of 30mg, 60mg and 120mg respectively, after randomization of patients.

Numerical congruity analysis, power sampling, biometric characteristics of internal compatibility between cohorts and outcome analysis with comparison for continuous homoscedastic case-control variables

Drafting of formal statistical analysis, drafting of information synopsis, writing, validation, forwarding to scientific journal and correction until obtaining, where possible, publications of the manuscript relating to the research.

ELIGIBILITY:
Inclusion Criteria: Hb<11; Having had Heart Surgery, Being Discharged to Rehab

-

Exclusion Criteria:

* Hb>11.1, hematological primary disesases

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-23 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 30 days
  Hemoglobin level at 30 day of treatment

SECONDARY OUTCOMES:
Martial Metabolism | 30 days
  Ferritin, Transferrin, Iron Saturation

CONTACTS AND LOCATIONS:
Overall Officials: Luca Paolo P Weltert, MD, Principal Investigator — European Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: One year after closure of study
Access Criteria: Reasonable Request

REFERENCES:
- [Background] Pierelli L, De Rosa A, Falco M, Papi E, Rondinelli MB, Turani F, Weltert L. Preoperative Sucrosomial Iron Supplementation Increases Haemoglobin and Reduces Transfusion Requirements in Elective Heart Surgery Patients: A Prospective Randomized Study. Surg Technol Int. 2021 Oct 28;39:321-328. doi: 10.52198/21.STI.39.CV1512. PMID 34710946
- [Background] Venturini E, Iannuzzo G, DI Lorenzo A, Cuomo G, D'Angelo A, Merone P, Cudemo G, Pacileo M, D'Andrea A, Vigorito C, Giallauria F. Short-term treatment of iron deficiency anemia after cardiac surgery. Int J Cardiol Heart Vasc. 2022 May 2;40:101038. doi: 10.1016/j.ijcha.2022.101038. eCollection 2022 Jun. PMID 35514874
- [Background] Weltert LP, De Rosa A, Rondinelli MB, Falco M, Turani F, Pierelli L. Benefits of pre-operative oral Sucrosomial(R) iron supplementation in cardiac surgery: influence of patient's baseline hemoglobin and gender. Blood Transfus. 2023 Jul;21(4):305-313. doi: 10.2450/2022.0222-22. Epub 2022 Nov 25. PMID 36580029